CLINICAL TRIAL: NCT05963256
Title: Investigation for Development of Predictive Model for Train of Four (TOF)% for Neurophysiological Monitoring During Neuroanesthesia
Brief Title: Prediction Model for TOF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eunah Cho, MD (Other)
Responsible Party: Sponsor-Investigator, Eunah Cho, MD, Assistant Professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Other Study IDs: 2023-01-056
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Neurophysiologic Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Twitch Electrode Array — Monitor train-of-four (TOF) count and percentage

SUMMARY:
This study was aimed to investigate a prediction model for predicting train-of-four (TOF) 50% in patients undergoing neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing neurosurgery
* scheduled for intra-operative neurophysiological monitoring
* American Society of Anesthesiologists physical class I, II, III

Exclusion Criteria:

* unable to monitor train-of-four
* decline to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing neurosurgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Train-of-four (TOF) ratio | 30 minutes after reaching the TOF plateau
  The ratio of the height of the fourth muscle response to the first one following the nerve stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, PhD, Principal Investigator — KangbukSamsung Hospital
Locations (1):
- Eunah Cho, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided